CLINICAL TRIAL: NCT03537677
Title: Sit Less for Successful Aging: A Sedentary Behavior Intervention for Older Adults in Independent Living Communities
Brief Title: Sit Less for Successful Aging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Andrea Hergenroeder, Assistant Professor, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17020397
Record Dates: First submitted 2018-05-15; First posted 2018-05-25 (Actual); Last update posted 2018-05-25 (Actual); Status verified 2018-05

CONDITIONS: Sedentary Lifestyle
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sedentary Behavior Intervention (Experimental): A behavioral intervention that targets prolonged sitting and encourages frequent activity breaks.
  Interventions: Behavioral: Reduction in Sedentary Behavior

INTERVENTIONS:
Behavioral: Reduction in Sedentary Behavior — This 12-week intervention targets a reduction in prolonged sitting and includes provision of a wrist-worn activity prompter and in-person group sessions with behavioral counseling.

SUMMARY:
The objective of this pilot study is to quantify patterns of activity and sedentary behavior in independent living residents and to collect preliminary data on the feasibility of reducing sedentary behavior using a 12-week, behavioral intervention in older adults. We will also measure the effects of reducing sedentary behavior on physical function, sleep, quality of life, energy/mood, pain and blood pressure. Participants will act as their own controls through the use of a double baseline period to examine stability of the physical activity and outcome measures.

DETAILED DESCRIPTION:
Aim 1: To measure the amount of sedentary time and ambulation (steps) in older adults residing in independent living communities.

Aim 2: To test the acceptability and effectiveness of a 12-week sedentary behavior intervention to decrease sitting and increase ambulation which will in turn improve physical function (primary outcome) as well as sleep, quality of life, energy/mood, pain and blood pressure (secondary outcomes) in independent living residents.

Background: Sedentary behavior, or sitting for prolonged periods during waking time, is identified as a health risk that is distinct from the failure to achieve sufficient physical activity. Older adults exhibit the greatest time in sedentary behavior which is concerning given its association with chronic disease and poorer physical function. Preliminary data suggest that individuals in long term care facilities may have even greater sedentary time due to personal factors and environment influences. Most often, exercise is targeted as a mechanism for ameliorating frailty in older adults; however, reduction in sedentary time may be a more appealing and realistic goal for improving health outcomes. Despite this, studies targeting sedentary time in older adults, particularly in those in independent living facilities, are lacking.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60 years
* Reside in an independent living facility
* Ability to walk approximately 100 feet (length of a hallway) with or without an assistive device

Exclusion Criteria:

* Unable to provide informed consent
* Presence of a comorbid medical condition that would limit ability to stand and perform light activity (e.g. recent orthopedic injury/surgery involving the lower extremities, currently undergoing treatment for cancer,acute cardiovascular conditions)
* Presence of a skin condition that would prohibit the use of an activity device attached with medical tape to the thigh (e.g. open wound on the thigh, skin infection on the lower extremity)

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-05-09 (Actual); Primary Completion 2017-10-03 (Actual); Study Completion 2017-10-03 (Actual)

PRIMARY OUTCOMES:
Change in Sedentary Behavior | Baseline to 12 weeks
  Objectively measured minutes of sitting during waking hours measured using the ActivPAL physical activity monitor for a minimum of 5 days pre and post-intervention. The ActivPAL is a thigh-mounted, compact device that classifies an individual's free-living activity into time spent in sedentary, standing, and walking behaviors.
Steps per Day | Baseline to 12 weeks
  The number of steps per day measured using the ActivPAL activity monitor. This monitor is worn for a minimum of 5 days before and after the intervention.
Short Physical Performance Battery | Baseline to 12 weeks
  This performance-based measure of physical function is a battery of measures to assess standing balance, gait speed and lower extremity strength (time to complete five chair rises)
Patient Reported Outcomes Measurement Information System (PROMIS) Physical Function Short Form 10a | Baseline to 12 weeks
  This self-report measure of physical function has 10 questions that assess the ability to perform various activities that require physical capability.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea L Hergenroeder, PT, PhD, Principal Investigator — Assistant Professor, Department of Physical Therapy
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No